CLINICAL TRIAL: NCT03717675
Title: A Prospective, Multi-Center, Non-randomized, Single Arm, Open Label, Supplemental Study to Evaluate the Safety and Effectiveness of the NovaCross™ Micro-catheter in Facilitating Crossing Chronic Total Occlusion (CTO) Coronary Lesions
Brief Title: Supplemental Study to Evaluate the Safety and Effectiveness of the NovaCross™ Micro-catheter
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nitiloop Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NT-CLP-03
Record Dates: First submitted 2018-10-21; First posted 2018-10-24 (Actual); Last update posted 2019-12-03 (Actual); Status verified 2019-12

CONDITIONS: Coronary Occlusion
MeSH Terms: conditions — Coronary Occlusion

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Interventional (Experimental): Interventional arm, where the NovaCross™ CTO micro-catheter will be placed in study subjects during the Total Occlusion opening procedure.
  Interventions: Device: NovaCross™ Chronic Total Occlusion micro-catheter

INTERVENTIONS:
Device: NovaCross™ Chronic Total Occlusion micro-catheter — The NovaCross™ micro catheter is a guidewire positioning and support micro catheter for improving chronic total occlusion (CTO) crossability. The NovaCross™ gains its supportive characteristics through the use of a unique operator-controlled Nitinol scaffold and an extendable segment. Investigators will use the NovaCross Micro catheter during a standard of care catheterization of patients diagnosed with coronary total occlusion.

SUMMARY:
This study will include up to 60 eligible male and female subjects. The purpose of this trial is to evaluate the safety and effectiveness of the NovaCross™ micro-catheter when used to facilitate crossing of Chronic Total Occlusion (CTO) lesions in coronary arteries. The procedure will be conducted on consenting patients diagnosed with a CTO in a coronary vessel that requires revascularization after a previously failed attempt to cross or refractory to 10 minutes of conventional guidewire attempt. This study is an extension study of Nitiloop's Pivotal study.

DETAILED DESCRIPTION:
The purpose of this trial is to evaluate the safety and effectiveness of the NovaCross™ micro-catheter when used to facilitate crossing of Chronic Total Occlusion (CTO) lesions in coronary arteries. The procedure will be conducted on consenting patients diagnosed with a CTO in a coronary vessel that requires revascularization after a previously failed attempt to cross or refractory to 10 minutes of conventional guidewire attempt.

ELIGIBILITY:
Inclusion Criteria:

1. Adult aged 25-80
2. Patient understands and has signed the study informed consent form
3. Patient has an angiographic documented Chronic Total Occlusion (i.e. >3 months occlusion duration) showing distal TIMI flow 0, with a reference diameter of at least 2 millimeters.
4. Left ventricle ejection fraction > 25%

Exclusion Criteria:

1. Patient unable to give informed consent. 2. Elevated CK-MB or troponin at baseline 3. Patient is known or suspected not to tolerate the contrast agent 4. Chronic Total Occlusion is located in aorto-ostial location, SVG CTO, in-stent occlusion 5. Appearance of a fresh thrombus or intraluminal filling defects 6. Intolerance to Aspirin and/or inability to tolerate a second antiplatelet agent (Clopidogrel and Prasugrel and Ticagrelor) 7. Cardiac intervention within 4 weeks of the procedure 8. Severe renal insufficiency with eGFR<30 ml/min/1.72 m2 9. Congestive heart failure [New York Heart Association (NYHA) Class III\IV] CSA Class IV 10. Life expectancy < 2 years due to other illnesses 11. Acute or unstable medical disorder/disease that may cause a risk to patient, including: i. Recent myocardial infarction (MI) (within the past two weeks) ii. Significant anemia (e.g. hemoglobin < 8.0 mg / dl) iii. Recent major cerebrovascular event (history of stroke or TIA within 1 month) iv. Severe uncontrolled systemic hypertension (e.g., >180/100 mmHg) v. Unstable angina requiring emergent percutaneous trans-luminal coronary angioplasty (PTCA) or coronary artery bypass graft (CABG)

Ages: 25 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2018-10-01 (Actual); Primary Completion 2019-07-17 (Actual); Study Completion 2019-11-01 (Actual)

PRIMARY OUTCOMES:
Primary Safety Endpoint - Rate of In hospital MACE events | until discharge or 30 days, the sooner of the two
  defined as the composite of death, myocardial infarction (MI), or urgent revascularization (target vessel revascularization (TVR) or urgent coronary artery bypass surgery (CABG)).
Primary Efficacy Endpoint - Intra-procedural technical success | during the procedure
  defined as the ability of the NovaCross™ microcatheter to successfully facilitate placement of a guidewire beyond a native coronary chronic total occlusion (CTO) in the true vessel lumen

SECONDARY OUTCOMES:
Rate of Lesion Crossing | during the procedure
  The ability to cross the lesion with a guidewire in the true lumen, effectively dilate the CTO lesion, and place a coronary stent with residual lumen stenosis of less than 30% while restoring antegrade TIMI 3 flow
Guidewire Facilitation and rate of successful penetration to the CTO | during the procedure
  The ability of the NovaCross™ micro-catheter to facilitate a guidewire successfully penetrating the proximal cap of the CTO
Crossability | during the procedure
  The effectiveness of the extendable portion in intra-CTO microcatheter crossability
Investigator visualization and ease of use | during the procedure
  The ability to have full visualization of the NovaCross during the CTO procedure and assessing the usability of the device
Myocardial Infraction (MI) Rate | up to 30 days
  In hospital MI rate
Device Related Adverse Events | up to 30 days
  Device-related perforation at the site of target coronary lesion and/or its proximal reference segment

CONTACTS AND LOCATIONS:
Overall Officials: Simon Walsh, MD, Principal Investigator — Belfast Health and Social Care Trust
Locations (3):
- Rabin Medical Center, Petah Tikva, Israel
- Samodzielny Publiczny Zakład Opieki Zdrowotnej Szpital Uniwersytecki w Krakowie, Krakow, Poland
- Belfast City Hospital, Belfast, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided